CLINICAL TRIAL: NCT07385820
Title: An Interventional Study Evaluating Two Different School Deployment Strategies, Testing the Effects of Onsite Awareness Raising on the Adoption of the Fruit-stands by Local Student Populations
Brief Title: A Comparative Intervention Study on Strategies for Fruit Distribution and Awareness Campaigns in Schools
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ioannis Ioakeimidis, Senior Researcher, Research Team Leader, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dnr 2024-07536-01; 101104618 - PREVENT (Other Grant/Funding Number: European Commission: European Health and Digital Executive Agency (HADEA))
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Dietary Behaviors; Fruit Consumption; Dietary Habits; Healthy Eating; Health Promotion; Schools
Keywords: Healthy eating; Dietary behavior; Fruit consumption; School environment; School; Health promotion; Prevention; Behavior change; Implementation study; School-based intervention; Public health; Adolescent health
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruit stands only (Experimental): Schools assigned to this arm receive fruit stands that provide free fruit during the school day. No awareness or educational campaign is implemented. Students report all their meals including fruits and snacks using the research mobile app before, during, and after the intervention
  Interventions: Behavioral: Fruit Stand Availability
- Fruit stands + awareness campaign (Experimental): Schools assigned to this arm receive fruit stands identical to the fruit-only arm, plus a school-based awareness campaign designed to promote healthy eating and encourage fruit consumption. Students report all their meals including fruits and snacks using the research mobile app before, during, and after the intervention.
  Interventions: Behavioral: Fruit Stand Availability; Behavioral: Awareness Campaign

INTERVENTIONS:
Behavioral: Fruit Stand Availability — Free fruit is provided to students through fruit stands placed in central school areas. Two fruit varieties are offered, and fruit uptake is monitored using digital scales integrated into the stands. Students photograph school-provided fruit before eating it and annotate it as "school fruit" in the app, while also documenting all meals and snacks as part of the study protocol.
Behavioral: Awareness Campaign — A school-based awareness campaign is delivered to promote healthy eating and encourage fruit consumption. Activities may include posters, messaging, or informational content. The campaign is implemented alongside the fruit stands to enhance student engagement with the intervention.
  Arms: Fruit stands + awareness campaign

SUMMARY:
This implementation study evaluates two strategies to increase fruit consumption among Swedish students. (1) installing fruit stands in schools and (2) combining fruit stands with a health-awareness campaign. The intervention is implemented in a set of participating schools, each following one of the predefined strategies. Students are asked to use a research app to photograph their meals and snacks during three data-collection periods before, during, and after the intervention. The study collects information on fruit intake, eating patterns, and the number of fruits taken from the stands to assess effectiveness and reduce food waste. The aim is to identify which strategy better supports healthy eating habits in school environments.

DETAILED DESCRIPTION:
This study is part of the Europe (EU) project "Improving and upscaling primary prevention of cancer by addressing childhood obesity through implementation research" (PREVENT), which aims to promote healthier dietary habits among students by improving access to fruits in school environments. The intervention is implemented in a set of participating schools, each assigned to one of the predefined strategies. The study examines whether providing fruit ad libitum during school hours influences students' snacking patterns, and whether an accompanying awareness campaign adds value beyond fruit availability alone.

In each participating school, fruit stands offering two types of fruit will be placed in central areas where students typically gather. Fruit will be available during periods when students have access to common spaces, and digital scales integrated into the stands will enable weight-based monitoring of fruit uptake. Designated school staff will photograph scale readings at the beginning, end, and one or more intermediate points during the day. These images will be processed using optical character recognition (OCR) to extract weight data and upload it to a secure backend system for automated monitoring of fruit distribution and potential food waste.

To evaluate students' eating behaviour and fruit consumption patterns, participating students will use a research mobile application to photograph their meals and snacks. Data collection takes place in three periods: (1) a baseline period prior to the introduction of fruit stands, (2) an early-intervention period immediately following the introduction of the stands, during which students continue to report all meals to capture short-term behavioural changes, and (3) a post-intervention period to assess sustained effects. The app records time and location metadata for each entry, allowing analysis of when and where food is consumed and how eating patterns change during the intervention.

The primary aim is to assess whether increased availability of free fruit influences students' snacking habits and whether the addition of an awareness campaign further enhances engagement with the fruit stands. Secondary aims include evaluating the feasibility of weight-based digital monitoring, characterising patterns of fruit uptake over the school day, and examining changes in students' overall eating behaviour across measurement periods. All data will be analysed at group level, and the study is considered minimal risk. Findings will support future scalable strategies for fruit distribution in school settings and contribute to broader evaluation of school-based dietary promotion initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in a Swedish school (elementary, middle, or high school)
* Ages 7-19 years
* Able to use a mobile phone to document meals and snacks
* Provided informed consent (with parental consent required for participants under 15 years old)

Exclusion Criteria:

- Presence of any clinically significant disease or condition that, in the opinion of the research team, may interfere with participation or influence study outcomes

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in fruit consumption | From enrollment until the end of Post-measurements (10 weeks after enrollment)
  Measured across baseline, early-intervention, and follow-up to evaluate whether fruit consumption differs between schools receiving fruit stands alone and those receiving fruit stands plus an awareness campaign.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Internationella Engelska Gymnasiet Södermalm, Stockholm
  - Blackebergs gymnasium, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share anonymized individual participant data (IPD) in accordance with our ethical approval. Fully anonymous subsets of the data may be made available to external researchers, including through open data repositories, if permitted under the ethical approval and the EU Open Data Directive. External access to anonymized IPD will be considered upon reasonable request and subject to compliance with ethical, legal, and data protection rules."